CLINICAL TRIAL: NCT05802030
Title: Effects of Plyometric Training on Physical Fitness and Serve Performance Among University Female Tennis Players
Brief Title: Effects of Plyometric Training on University Female Tennis Players' Physical Fitness and Serve Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Deng Nuannuan, PHD candidate, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Deng Nuannuan
Record Dates: First submitted 2023-03-03; First posted 2023-04-06 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Physical Illness; Skill, Coping
Keywords: Physical fitness; Serve performance; Plyometric training
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric training (Experimental): The 8 weeks of plyometric training included push-ups and medicine ball exercises for the upper limbs and jumping, hopping exercises for the lower limbs. Exercises for the upper limbs were immediately followed by lower-limb exercises, with no intervening rest periods.
  Interventions: Other: Plyometric training
- Routine training (Active Comparator): During the intervention, the control group just continued with their routine training regime (e.g., normal fitness training, and injury prevention drills), twice a week, for the duration of the experiment.
  Interventions: Other: Routine training

INTERVENTIONS:
Other: Plyometric training — Plyometric training can be described as a type of exercise that involves a rapid and forceful movement that consists of an eccentric contraction, followed by an immediate and explosive concentric contraction. Upper and lower limb plyometrics are exercises that enable an upper and lower body muscle group to react quickly to produce maximal strength
  Arms: Plyometric training
Other: Routine training — Regular tennis training, including normal fitness training, and injury prevention drills
  Arms: Routine training

SUMMARY:
The main objective of this study is to examine the effects of upper and lower limb plyometric training on the selected physical fitness and serve performance among university female tennis players in China.

The main hypothesis of this study is to evaluate whether there are significant effects of 8 weeks of upper and lower limb plyometric training on selected physical fitness and serve performance among university female tennis players in China.

DETAILED DESCRIPTION:
This intervention lasted for 8 weeks, two times each week, for 30-60 minutes of low-high intensity exercise. The content of the experimental group and control group of exercises mainly includes warm-up, primary content, and cool down. The intervention included push-ups and medicine ball exercises for the upper limbs and jumping, hopping exercises for the lower limbs. Exercises for the upper limbs were immediately followed by lower-limb exercises, with no intervening rest periods. all plyometric exercises, including those involving the upper and lower limbs, were executed with maximal effort, with the goal of reducing contact time during each repetition, and with no allowance for rest periods between jumps. During the intervention, the control group just continued with their regular training regime (e.g., normal fitness training, and injury prevention drills), twice a week, for the duration of the experiment.

ELIGIBILITY:
Inclusion Criteria:

1. University female tennis players (aged 18-24 years old);
2. Players who had been trained professionally for more than three years
3. No history of recent surgery, no rehabilitation for the past 12 months;
4. Not systematically trained in plyometric training;

Exclusion Criteria:

1. Tennis-specific training time less than 3 years;
2. Players with a history of recent fractures or any injury;
3. Presently involved in a plyometric training program;

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-08 (Actual); Primary Completion 2023-06-18 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline power performance at 4 weeks and 8 weeks | Pretest: Before experiment; Mid-test: 4 weeks end; Post-test: 8 weeks end
  Power is the ability to perform strength based movements quickly.
Change from baseline strength performance at 4 weeks and 8 weeks | Pretest: Before experiment; Mid-test: 4 weeks end; Post-test: 8 weeks end
  Strength is the maximal force or torque that a muscle can generate.
Change from baseline speed performance at 4 weeks and 8 weeks | Pretest: Before experiment; Mid-test: 4 weeks end; Post-test: 8 weeks end
  The ability to move all or part of the body as quickly as possible
Change from baseline agility performance at 4 weeks and 8 weeks | Pretest: Before experiment; Mid-test: 4 weeks end; Post-test: 8 weeks end
  Agility is a skill considered to be important for many sports and has been defined as "a rapid whole-body movement with change of velocity or direction in response to a stimulus.
Change from baseline endurance performance at 4 weeks and 8 weeks | Pretest: Before experiment; Mid-test: 4 weeks end; Post-test: 8 weeks end
  Endurance describes your body's ability to maintain physical activity for an extended amount of time.
Change from baseline flexibility performance at 4 weeks and 8 weeks | Pretest: Before experiment; Mid-test: 4 weeks end; Post-test: 8 weeks end
  Flexibility is the ability to move muscles and joints through a full normal range of motion.
Change from baseline serve velocity performance at 4 weeks and 8 weeks | Pretest: Before experiment; Mid-test: 4 weeks end; Post-test: 8 weeks end
  It is one of the most repeated strokes during the game.
Change from baseline serve accuracy performance at 4 weeks and 8 weeks | Pretest: Before experiment; Mid-test: 4 weeks end; Post-test: 8 weeks end
  In many sports, the accuracy of the execution of a motor skill determines success or failure.

CONTACTS AND LOCATIONS:
Overall Officials: Nuannuan Deng, Principal Investigator — Universiti Putra Malaysia
Locations (2):
- China (2):
  - Chongqing university, Chongqing
  - Southwest university, Chongqing

IPD SHARING:
Plan to Share IPD: No
Since this is my doctoral thesis experiment, I won't share it until I graduate

REFERENCES:
- [Background] Deng N, Soh KG, Zaremohzzabieh Z, Abdullah B, Salleh KM, Huang D. Effects of Combined Upper and Lower Limb Plyometric Training Interventions on Physical Fitness in Athletes: A Systematic Review with Meta-Analysis. Int J Environ Res Public Health. 2022 Dec 28;20(1):482. doi: 10.3390/ijerph20010482. PMID 36612806
- [Background] Fernandez-Fernandez J, Saez de Villarreal E, Sanz-Rivas D, Moya M. The Effects of 8-Week Plyometric Training on Physical Performance in Young Tennis Players. Pediatr Exerc Sci. 2016 Feb;28(1):77-86. doi: 10.1123/pes.2015-0019. Epub 2015 Aug 6. PMID 26252503
- [Background] Elliott B. Biomechanics and tennis. Br J Sports Med. 2006 May;40(5):392-6. doi: 10.1136/bjsm.2005.023150. PMID 16632567